CLINICAL TRIAL: NCT01066130
Title: Psychosocial Treatment Intervention in Persons Newly Diagnosed With Rheumatoid Arthritis or Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Norrbacka-Eugenia Foundation (Other); Swedish Rheumatism Foundation (Unknown); Svenska Diabetes Association (Unknown)
Responsible Party: Catharina Gafvels, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KI DNR 00-065; Other Grant/Funding Number (Other Grant/Funding Number: Norrbacka-Eugeniastiftelsen 811/06); Other Grant/Funding Number (Other Grant/Funding Number: Reumatikerfonden D:nr 45/05)
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Diabetes Mellitus; Arthritis, Rheumatoid; Coping Skills
Keywords: Diabetes Mellitus; Arthritis, Rheumatoid; psychosocial aspects; Patient Adherence; Social Work; Coping Behavior; Coping Skills; Adaptation, Psychological
MeSH Terms: conditions — Diabetes Mellitus; Arthritis, Rheumatoid; Patient Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intensive treatment arm (Experimental): Every second person with psychosocial problems was randomized into this arm. The intervention consisted of personalized, intensive psychosocial treatment provided by a medical social worker on the basis of the patient's problems for up to 2 years after inclusion.
  Interventions: Behavioral: Intensive individualized psychosocial treatment
- Minimal treatment arm (Experimental): Every second patient with psychosocial problems was assigned to this arm. Patients in this arm received minimal social support by a medical social worker.
  Interventions: Behavioral: Minimal treatment arm
- No need for psychosocial treatment (No Intervention): This arm consisted of individuals who did not need psychosocial treatment or measures. The need for such treatment and measures was determined at baseline for all persons included in the study.

INTERVENTIONS:
Behavioral: Intensive individualized psychosocial treatment — Each person was given psychosocial treatment and support by a medical social worker a maximum of one time each week for a period of up to 2 years after inclusion. Treatment was designed by a medical social work on the basis of the individual's personal needs.
  Arms: Intensive treatment arm
Behavioral: Minimal treatment arm — Minimal social measures were provided to individuals in this arm. No treatment that included conversational therapy was given.
  Arms: Minimal treatment arm

SUMMARY:
The aim of this study is to evaluate the results of psychosocial treatment in patients with newly diagnosed rheumatoid arthritis and/or diabetes.

DETAILED DESCRIPTION:
Research and clinical experience show that adaptation to chronic disease is affected by individuals' psychological and social situations and subjective experiences of threat to identity, autonomy, and life. It is important to identify persons whose psychosocial situation and reaction to the diagnosis is such that they may not be able to adjust to the illness or take adequate responsibility for adherence to treatment.

The purpose of this study is to identify such at-risk persons, and with the help of psychosocial treatment, strengthen their resistance resources and help them work through emotional and social problems that hinder adequate adaptation and adherence to treatment.

Beginning in 2001, 200 consecutive patients between 18 and 65 years who are newly diagnosed with either rheumatoid arthritis (n = 100) or diabetes (n = 100) at the Karolinska Hospital, Solna, Sweden, will be included in the study. Each person will be interviewed by a medical social worker about their psychosocial situation and possible problems. Every other patient with psychosocial problems will be offered intensive, personalized psychosocial treatment. The rest of the patients with problems will be given minimal required measures. The psychosocial well-being and medical situation of all patients (intensive treatment group, minimal treatment group, and the group without need of psychosocial measures) will be followed for 2 years and evaluated at the conclusion of that time.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed diabetes (within one month of receiving diagnosis)
* newly diagnosed rheumatoid arthritis(within one month of receiving diagnosis)
* patient at the endocrinological or rheumatical clinic at the Karolinska University Hospital, Solna, Sweden

Exclusion Criteria:

* patients previously diagnosed with diabetes (had been diagnosed more than a month ago)
* patients previously diagnosed with rheumatoid arthritis (had been diagnosed more than a month ago)
* inability to speak Swedish well enough to fill in standard questionnaires

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2001-01; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Psychosocial well-being as measured by interview with a medical social worker, Hospital Anxiety and Depression Scale, General Coping Questionnaire, Social Situation Questionnaire, and self-reported satisfaction with psychosocial treatment | 2 years after inclusion

SECONDARY OUTCOMES:
Medical parameters that show whether the patient has reached treatment goals for his or her disease; for example, glycated hemoglobin (HbA1c) for diabetes and the Disease Activity Score (DAS) for rheumatoid arthritis | 2 years after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Catharina M Gafvels, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Center for Family and Community Medicine, Huddinge
  - Karolinska University Hospital Solna, Stockholm